CLINICAL TRIAL: NCT01530685
Title: Effect of Glycabiane, a Dietary Supplement, on Glycemic Control of Prediabetic Subjects
Brief Title: Gycabiane and Glycemic Control of Prediabetic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PiLeJe (Industry)
Responsible Party: Sponsor
Organization: Larena SAS (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PILEJE-Glyca-0910
Record Dates: First submitted 2011-12-05; First posted 2012-02-10 (Estimated); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Hyperglycemia
Keywords: cinnamon; chromium; prediabete; overweight
MeSH Terms: conditions — Hyperglycemia; Overweight | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glycabiane, gelule (Experimental)
  Interventions: Dietary Supplement: Glycabiane
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Glycabiane — 2 gelule per day for 4 months
  Other Names: Dietary supplement
  Arms: Glycabiane, gelule
Dietary Supplement: placebo — 2 gelules per day for 4 months
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effects of supplementation Glycabiane, a dietary supplement, on glycemic control of overweight prediabetic subjects.

DETAILED DESCRIPTION:
Cinnamon's effects on blood glucose have been the subject of many clinical and animal studies; however, the issue of cinnamon intake's effect on fasting blood glucose (FBG) in people with prediabetes still remains unclear.

The main purpose of this study is to examine the effects of supplementation with Glycabiane, a dietary supplement rich in cinnamon extract, on fast blood glucose of overweight prediabetic subjects in a randomized, placebo-controlled, clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female from 25 to 65 years old
* 1.0g/L ≤ fast blood glucose < 1.26g/L
* overweight (IMC > 25)

Exclusion Criteria:

* thyroid disease
* hypogonadism
* History of musculoskeletal, autoimmune or neurological disease
* Treatment against thyroid disease, hypoglycemia, hypertension, or anti-coagulant
* Pregnant or lactating women

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2011-10-27 (Actual); Primary Completion 2012-09-25 (Actual); Study Completion 2012-09-25 (Actual)

PRIMARY OUTCOMES:
Fast Blood Glucose | 4 months
  Fast blood glucose will be measured before and after 4 months of supplementation and after 2 months of wash-out

CONTACTS AND LOCATIONS:
Overall Officials: Karine Clément, MD, Principal Investigator — INSERM U872
Locations (1):
- CHU Pitié Salpetriere, Paris, France

REFERENCES:
- [Derived] Liu Y, Cotillard A, Vatier C, Bastard JP, Fellahi S, Stevant M, Allatif O, Langlois C, Bieuvelet S, Brochot A, Guilbot A, Clement K, Rizkalla SW. A Dietary Supplement Containing Cinnamon, Chromium and Carnosine Decreases Fasting Plasma Glucose and Increases Lean Mass in Overweight or Obese Pre-Diabetic Subjects: A Randomized, Placebo-Controlled Trial. PLoS One. 2015 Sep 25;10(9):e0138646. doi: 10.1371/journal.pone.0138646. eCollection 2015. PMID 26406981